CLINICAL TRIAL: NCT00850135
Title: Correlation of Continuous Glucose Monitoring and Glucose Tolerance Testing With Pregnancy Outcomes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Yasser Yehia El-Sayed, Professor of Obstetrics and Gynecology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SU-02052009-1738; IRB #12335 (Other: Stanford University Medical Center IRB)
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes, Gestational
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Continuous Glucose Monitor in pregnancy (Other): The Seven Continuous Glucose Monitoring System: Between 24-28 weeks of gestation, the recommended period of glucola testing, a soft sensor for continuous glucose monitoring system (CGMS) will be inserted superficially under the skin. The patient will be instructed on how to wear and care for the device. She will wear the CGMS for 7 days, then return to the clinic for removal of the device, and downloading of the data. Finger stick blood glucoses will be checked by the patient 2 times daily during the 7 days of wearing the CGMS.
  Interventions: Device: The Seven Continuous Glucose Monitoring System

INTERVENTIONS:
Device: The Seven Continuous Glucose Monitoring System — Between 24-28 weeks of gestation, the recommended period of glucola testing, a soft sensor for continuous glucose monitoring system (CGMS) will be inserted superficially under the skin. The patient will be instructed on how to wear and care for the device. She will wear the CGMS for 7 days, then return to the clinic for removal of the device, and downloading of the data. Finger stick blood glucoses will be checked by the patient 2 times daily during the 7 days of wearing the CGMS.

SUMMARY:
Diabetic pregnant patients are at risk for adverse pregnancy outcomes, including larger than expected fetuses and unplanned operative deliveries, due to elevated blood glucose levels. the one-hour glucola test is currently used to screen pregnant patients for gestational diabetes. This involves ingesting a 50-gram glucose load, followed by a blood test one hour later. We wish to compare 7-day continuous glucose monitoring to the one-hour glucola test, and determine which one correlates better with adverse pregnancy outcomes as well as which one more accurately identifies patients at risk for adverse pregnancy outcomes.

DETAILED DESCRIPTION:
All pregnant patients without pre-existing diabetes will be eligible for the study. Interest in participation will be determined at their initial prenatal visit. Those that are interested will be consented. Between 24-28 weeks of gestation, the recommended period of glucola testing, a soft sensor for continuous glucose monitoring system (CGMS) will be inserted superficially under the skin. The patient will be instructed on how to wear and care for the device. She will wear the CGMS for 7 days, then return to the clinic for removal of the device, and downloading of the data. She will perform the routine glucola test sometime between days 2 to 7 . Finger stick blood glucoses will be checked by the patient 2 times daily during the 7 days of wearing the CGMS. Results of CGMS will not be available to the patient or her physician until after completion of the pregnancy. The patient will be treated routinely, based on the results of the routine glucola test.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients
* Age 18-50
* Gestational age less than 28 weeks

Exclusion Criteria:

* Minors less than 18 years of age
* Multiple gestation
* Known fetal anomalies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2009-02; Primary Completion 2014-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Yehia El-Sayed, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Santa Clara Valley Medical Center, San Jose, California
  - Stanford University School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sung JF, Kogut EA, Lee HC, Mannan JL, Navabi K, Taslimi MM, El-Sayed YY. Correlation of continuous glucose monitoring profiles with pregnancy outcomes in nondiabetic women. Am J Perinatol. 2015 Apr;32(5):461-8. doi: 10.1055/s-0034-1390344. Epub 2014 Sep 28. PMID 25262455

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Glucose Monitor for Diabetes in Pregnancy Screening: The Seven Continuous Glucose Monitoring System: Between 24-28 weeks of gestation, the recommended period of glucola testing, a soft sensor for continuous glucose monitoring system (CGMS) will be inserted superficially under the skin. The patient will be instructed on how to wear and care for the device. She will wear the CGMS for 7 days, then return to the clinic for removal of the device, and downloading of the data. Finger stick blood glucoses will be checked by the patient 2 times daily during the 7 days of wearing the CGMS.
Period: Overall Study
Arm/Group | Continuous Glucose Monitor for Diabetes in Pregnancy Screening
Started | 57
Completed | 56
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: A total of 57 patients were enrolled from two clinical sites. One patient had no CGM data. One patient transferred care after completing the CGM study period, and thus did not have delivery data. Two patients who had an existing diagnosis of diabetes were excluded.The remaining 53 patients were analyzed.
Arm/Group | Continuous Glucose Monitor for Diabetes in Pregnancy Screening
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 53
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 0
  White | 14
  More than one race | 2
  Unknown or Not Reported | 24
Region of Enrollment [Number; unit: participants]
  United States | 53
Gestational Age at Enrollment [Mean (Standard Deviation); unit: weeks] | 25.9 (1.2)
Parity [Number; unit: participants]
  Nulliparous | 23
  Multiparous | 30
Pre-pregnancy BMI [Mean (Standard Deviation); unit: kg/m2] | 29.1 (8.4)
BMI at enrollment [Mean (Standard Deviation); unit: kg/m2] | 32.5 (8.5)
Insurance status [Number; unit: participants]
  Public | 29
  Private | 24

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Glucose AUC and Birth Weight.
Description: For each patient's CGM data, we calculated the total area under the curve (AUC) for values above the predefined cutoffs of 110, 120, 130, 140, and 180 mg/dL. Patients wore the CGM for different amounts of time; therefore, the total AUC for the entire duration of CGM use was divided by the number of 24-hour periods of data collection. We called these normalized values "AUC-110," "AUC-120," "AUC-130," "AUC-140," and "AUC-180," and they reflect both the magnitude and duration of hyperglycemic excursions above the predetermined thresholds in an average 24-hour period. Birth weight percentile was determined using birth weight data derived from 1999 and 2000 United States Natality datasets. The correlation coefficient (r) was calculated between birth weight percentiles and each of the following: AUC-110, AUC-120, AUC-130, AUC-140, AUC-180, and 1-hour GCT result.
Time Frame: CGM measured 7 days at beginning of pregnancy,birth weight measured a time of delivery
Population: A total of 57 patients were enrolled from two clinical sites. Two patients did not have monitoring or delivery data.
  Two patients who had an existing diagnosis of diabetes were excluded. The remaining 53 patients were analyzed.
Measure: Number; unit: correlation coefficient
Arm/Group | Continuous Glucose Monitor for Diabetes in Pregnancy Screening
Number analyzed (Participants) | 53
correlation coefficient
  AUC-110 to birth weight centile | 0.2902
  AUC-120 to birth weight centile | 0.2935
  AUC-130 to birth weight centile | 0.2915
  AUC-140 to birth weight centile | 0.2859
  AUC-180 to birth weight centile | 0.2499
  1hr GCT to birth weight centile (n=44) | -0.0234
Statistical Analysis 1: Comparison: Continuous Glucose Monitor for Diabetes in Pregnancy Screening; Test type: Superiority or Other; p = 0.035, correlation — p-Value for the correlation between AUC-110 and birth weight

2. Secondary Outcome: Pregnancy and Delivery Characteristics for Participants With AUC-130 <= 22,000 and AUC-130 > 22,000
Description: For our secondary outcome analyses,we chose to focus on AUC-130 because 130 mg/dL is a common threshold used when treating gestational diabetics. In addition, 130 mg/dL was the threshold used in an earlier pilot study performed at our institution because it had the best correlation with birth weight percentile.
  Secondary outcomes were compared between these two groups using the chi-square test. Data were analyzed using Stata 11.2. AUC-130 values were divided into "high" and "low" at a cutoff of 22,000, which was the 90th percentile of AUC-130 values.
Time Frame: CGM measured 7 days at beginning of pregnancy,birth weight measured a time of delivery
Population: A total of 57 patients were enrolled from two clinical sites. Of these patients, 44 were screened with the 1-hour 50-g GCT; 9 were screened with 2-hour 75-g GTT. Complete data on secondary outcomes was available for 43 patients with 1-hour 50-g GCT and these were analyzed.
Measure: Number; unit: participants
Groups:
- Participants With AUC 130 <= 22,000; Participants With AUC 130 >22,000: AUC-130 values were divided into"high" and "low" at a cutoff of 22,000, which was the 90th percentile of AUC-130 values.
Arm/Group | Participants With AUC 130 <= 22,000 | Participants With AUC 130 >22,000
Number analyzed (Participants) | 38 | 5
participants
  Delivery Mode: Vaginal Delivery | 31 | 5
  Delivery Mode: Unplanned Operative Delivery | 7 | 0
  Macrosomia >90% | 4 | 1

ADVERSE EVENTS:
Arm/Group | Continuous Glucose Monitor for Diabetes in Pregnancy Screening
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

LIMITATIONS AND CAVEATS:
Limited monitoring period between 24 and 28 weeks' gestation. Sample size was under powered to detect differences in secondary outcomes of interest.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No